CLINICAL TRIAL: NCT04865029
Title: Acute Estradiol and Progesterone Therapy in Hospitalized Adults to Reduce Coronavirus Disease (COVID-19) Severity: A Randomized Control Trial
Brief Title: Estradiol and Progesterone in Hospitalized COVID-19 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment due to change of COVID 19 variant prevalence
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-939
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Estradiol; Progesterone; Covid19; Estrogen; Hormones; Progestogens; Depo-Estradiol; Prometrium; Micronized Progesterone
MeSH Terms: conditions — COVID-19 | interventions — estradiol 17 beta-cypionate; Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Standard of Care along with Estradiol Cypionate 5mg intramuscular injection at admission and Progesterone 200mg by mouth daily for 5 days starting at admission.
  Interventions: Drug: Estradiol Cypionate 5 mg/ml; Drug: Progesterone 200 mg Oral Capsule
- Control Arm (Other): Standard of Care along with placebo injection and placebo pill
  Standard of Care consistent with the National Institutes of Health (NIH) COVID-19 Treatment Guidelines
  Interventions: Other: Placebo injection and placebo pill

INTERVENTIONS:
Other: Placebo injection and placebo pill — Standard of Care consistent with the National Institutes of Health (NIH) COVID-19 Treatment Guidelines
  Arms: Control Arm
Drug: Estradiol Cypionate 5 mg/ml — Standard of Care along with Estradiol Cypionate 5mg intramuscular injection at admission.
  Arms: Treatment Arm
Drug: Progesterone 200 mg Oral Capsule — Standard of Care along with Progesterone 200mg by mouth daily for 5 days starting at admission.
  Arms: Treatment Arm

SUMMARY:
The purpose of this study is to determine to what extent a short systemic steroid therapy with estradiol and progesterone, administered early to hospitalized and confirmed COVID-19 positive patients of both sexes in addition to standard of care (SOC) can reduce the severity of symptoms and outcomes compared to SOC alone.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome Associated Corona Virus (SARS-CoV-2), causing COVID-19, has killed over 2.8 million people globally, including 550,000 in the US as of March 2021. Although, the vaccination campaign is ramping up, vaccination hesitancy in the United States represents up to 25-30% of the population, and hospitalizations and deaths are still at the level of 2020. Apart from corticosteroids, most available therapeutic options are at best marginally efficient in reducing disease severity and mortality and extremely expensive. Therefore, the systematic investigation of clinically approved drugs is a priority in order to determine what does improve the disease and invest resources to go to full-scale production. Our current understanding of the disease is that COVID-19 deaths result from an inappropriate immune response with outpouring of pro-inflammatory chemokines leading to lung infiltration and hyperactivation of monocytes and macrophages producing pro-inflammatory cytokines (cytokine storm), resulting in lung edema, reduced gas exchange, and ultimately leading to acute respiratory distress syndrome and multiorgan failure. Men with COVID-19 have a uniformly more severe outcome than women. In series from China, Europe and the U.S., COVID-19 mortality was consistently 1.5 to 2-fold higher in men than in women, suggesting that female biological sex is protecting women from COVID-19 mortality. It is established that women exhibit heightened immune responses to viral infections compared to men, which is at least partially due to the genetic benefit of gene dosage in X-linked immune-response genes. Ovarian steroids, however, also play a protective role. In New York City, among 5700 hospitalized patients, the female protection from COVID-19 mortality was observed at all ages, but was more pronounced in subjects under 50 years of age (18% mortality in women) compared to patients > 50 years of age (40.5% mortality in women), suggesting that ovarian steroids are involved in mitigating COVID-19 mortality in pre-menopausal women. Further, the analysis of electronic health records of over 68,000 COVID-19 patients revealed that estrogen therapy is associated with more than 50% reduction in mortality. The main female steroids, 17β-estradiol and progesterone exhibit potent immuno-modulatory and anti-inflammatory actions via estrogen and progesterone receptors expressed in all immune cells, including epithelial cells, macrophages, dendritic cells, cluster of differentiation 4 (CD4+) and cluster of differentiation 8 (CD8+) lymphocytes, and B cells. Progesterone also acts partially via the glucocorticoid receptor. Together estradiol and progesterone produce a state of decreased innate immune cells production of proinflammatory cytokines, enhanced T cells anti-inflammatory responses and immune tolerance, and enhanced B-cell-mediated antibody production. The National Institutes of Health (NIH) COVID-19 Treatment Guidelines Panel recommends the use of dexamethasone 6 mg per day for up to 10 days or until hospital Discharge (whichever comes first) as standard of care (SOC) for the treatment of hospitalized COVID-19 patients who require supplemental oxygen but who are not mechanically ventilated and for the treatment of hospitalized patients who are mechanically ventilated. Remdesivir is SOC at Tulane for COVID-19 patients who require supplemental oxygen but who are not mechanically ventilated. We believe that in hospitalized COVID-19 patients, a short treatment with the combination estradiol and progesterone, administered early and as a prevention in addition to SOC, will prevent or mitigate the cytokine storm while increasing antibody production and prevent severe outcomes, without side effects. Therefore, it will provide steroid immunomodulation without immunosuppression. The advantage of repurposing estradiol and progesterone compounds is the depth of knowledge regarding their clinical efficacy and toxicity that has accumulated from decades of clinical and basic studies. Estradiol and progesterone are widely available in hospitals, inexpensive, manufacturable to scale, and can be prescribed immediately.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization at Tulane Medical Center in the Department of General Internal Medicine and Geriatrics with COVID-19 (WHO Ordinal scale score 3-5) and confirmed by SARS-CoV-2 Polymerase Chain Reaction (PCR).
2. Respiratory symptoms (fever, shortness of breath or cough) or abnormal lung exam or chest imaging characteristic of mild to severe COVID-19 pneumonia.
3. Patient and/or legally authorized representative (LAR) agrees to comply with study procedures and the collection of blood samples per protocol.
4. Patient and/or LAR agrees to be placed on prophylactic dose of anticoagulation for prevention of deep venous thrombosis (DVT) (if necessary).
5. Patient or legally authorized representative has signed informed consent.
6. Women of childbearing age with a negative pregnancy test on admission.

Exclusion Criteria:

1. Patient under 18 years of age.
2. Critical COVID-19 (respiratory failure requiring intubation and mechanical ventilation, shock, multi-organ failure).
3. Pregnant women confirmed by pregnancy test.
4. Women who are within six weeks of postpartum.
5. Patient is not hospitalized at Tulane Medical Center with confirmed COVID-19.
6. Patient included in another COVID-19 trial (excluding hydroxychloroquine and dexamethasone).
7. Women already treated by estrogen and or progestogen therapy two weeks prior to admission.
8. Men already treated by testosterone therapy prior to admission.
9. History of breast or endometrial cancer.
10. Abnormal genital bleeding.
11. Active or recent (e.g., within the past year) stroke or myocardial infarction.
12. History of blood clots including deep vein thrombosis related to clotting disease, or pulmonary emboli (prior to hospitalization).
13. History of liver dysfunction or disease.
14. Patients with end-stage renal disease
15. Patients taking inhibitors of CYP3A4 such as erythromycin, clarithromycin, ketoconazole, itraconazole, and ritonavir.
16. Patients taking St. John's Wort preparations (Hypericum perforatum), phenobarbital, carbamazepine, and rifampin.
17. Patients within 6 weeks of major orthopedic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Mauvais-Jarvias, MD, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Blanco-Melo D, Nilsson-Payant BE, Liu WC, Uhl S, Hoagland D, Moller R, Jordan TX, Oishi K, Panis M, Sachs D, Wang TT, Schwartz RE, Lim JK, Albrecht RA, tenOever BR. Imbalanced Host Response to SARS-CoV-2 Drives Development of COVID-19. Cell. 2020 May 28;181(5):1036-1045.e9. doi: 10.1016/j.cell.2020.04.026. Epub 2020 May 15. PMID 32416070
- [Background] Chousterman BG, Swirski FK, Weber GF. Cytokine storm and sepsis disease pathogenesis. Semin Immunopathol. 2017 Jul;39(5):517-528. doi: 10.1007/s00281-017-0639-8. Epub 2017 May 29. PMID 28555385
- [Background] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Background] Tanaka T, Narazaki M, Kishimoto T. Immunotherapeutic implications of IL-6 blockade for cytokine storm. Immunotherapy. 2016 Jul;8(8):959-70. doi: 10.2217/imt-2016-0020. PMID 27381687
- [Background] McGonagle D, Sharif K, O'Regan A, Bridgewood C. The Role of Cytokines including Interleukin-6 in COVID-19 induced Pneumonia and Macrophage Activation Syndrome-Like Disease. Autoimmun Rev. 2020 Jun;19(6):102537. doi: 10.1016/j.autrev.2020.102537. Epub 2020 Apr 3. PMID 32251717
- [Background] Mauvais-Jarvis F, Bairey Merz N, Barnes PJ, Brinton RD, Carrero JJ, DeMeo DL, De Vries GJ, Epperson CN, Govindan R, Klein SL, Lonardo A, Maki PM, McCullough LD, Regitz-Zagrosek V, Regensteiner JG, Rubin JB, Sandberg K, Suzuki A. Sex and gender: modifiers of health, disease, and medicine. Lancet. 2020 Aug 22;396(10250):565-582. doi: 10.1016/S0140-6736(20)31561-0. PMID 32828189
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Klein SL, Dhakal S, Ursin RL, Deshpande S, Sandberg K, Mauvais-Jarvis F. Biological sex impacts COVID-19 outcomes. PLoS Pathog. 2020 Jun 22;16(6):e1008570. doi: 10.1371/journal.ppat.1008570. eCollection 2020 Jun. PMID 32569293
- [Background] Klein SL, Flanagan KL. Sex differences in immune responses. Nat Rev Immunol. 2016 Oct;16(10):626-38. doi: 10.1038/nri.2016.90. Epub 2016 Aug 22. PMID 27546235
- [Background] Phiel KL, Henderson RA, Adelman SJ, Elloso MM. Differential estrogen receptor gene expression in human peripheral blood mononuclear cell populations. Immunol Lett. 2005 Feb 15;97(1):107-13. doi: 10.1016/j.imlet.2004.10.007. PMID 15626482
- [Background] Straub RH. The complex role of estrogens in inflammation. Endocr Rev. 2007 Aug;28(5):521-74. doi: 10.1210/er.2007-0001. Epub 2007 Jul 19. PMID 17640948
- [Background] Mauvais-Jarvis F, Klein SL, Levin ER. Estradiol, Progesterone, Immunomodulation, and COVID-19 Outcomes. Endocrinology. 2020 Sep 1;161(9):bqaa127. doi: 10.1210/endocr/bqaa127. PMID 32730568
- [Background] Mauvais-Jarvis F, Manson JE, Stevenson JC, Fonseca VA. Menopausal Hormone Therapy and Type 2 Diabetes Prevention: Evidence, Mechanisms, and Clinical Implications. Endocr Rev. 2017 Jun 1;38(3):173-188. doi: 10.1210/er.2016-1146. PMID 28323934
- [Background] Mauvais-Jarvis F. Aging, Male Sex, Obesity, and Metabolic Inflammation Create the Perfect Storm for COVID-19. Diabetes. 2020 Sep;69(9):1857-1863. doi: 10.2337/dbi19-0023. Epub 2020 Jul 15. PMID 32669390
- [Background] Seeland U, Coluzzi F, Simmaco M, Mura C, Bourne PE, Heiland M, Preissner R, Preissner S. Evidence for treatment with estradiol for women with SARS-CoV-2 infection. BMC Med. 2020 Nov 25;18(1):369. doi: 10.1186/s12916-020-01851-z. PMID 33234138
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Khubchandani J, Sharma S, Price JH, Wiblishauser MJ, Sharma M, Webb FJ. COVID-19 Vaccination Hesitancy in the United States: A Rapid National Assessment. J Community Health. 2021 Apr;46(2):270-277. doi: 10.1007/s10900-020-00958-x. Epub 2021 Jan 3. PMID 33389421
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Kaka AS, MacDonald R, Greer N, Vela K, Duan-Porter W, Obley A, Wilt TJ. Major Update: Remdesivir for Adults With COVID-19 : A Living Systematic Review and Meta-analysis for the American College of Physicians Practice Points. Ann Intern Med. 2021 May;174(5):663-672. doi: 10.7326/M20-8148. Epub 2021 Feb 9. PMID 33560863
- [Background] Salvarani C, Dolci G, Massari M, Merlo DF, Cavuto S, Savoldi L, Bruzzi P, Boni F, Braglia L, Turra C, Ballerini PF, Sciascia R, Zammarchi L, Para O, Scotton PG, Inojosa WO, Ravagnani V, Salerno ND, Sainaghi PP, Brignone A, Codeluppi M, Teopompi E, Milesi M, Bertomoro P, Claudio N, Salio M, Falcone M, Cenderello G, Donghi L, Del Bono V, Colombelli PL, Angheben A, Passaro A, Secondo G, Pascale R, Piazza I, Facciolongo N, Costantini M; RCT-TCZ-COVID-19 Study Group. Effect of Tocilizumab vs Standard Care on Clinical Worsening in Patients Hospitalized With COVID-19 Pneumonia: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jan 1;181(1):24-31. doi: 10.1001/jamainternmed.2020.6615. PMID 33080005
- [Background] Janiaud P, Axfors C, Schmitt AM, Gloy V, Ebrahimi F, Hepprich M, Smith ER, Haber NA, Khanna N, Moher D, Goodman SN, Ioannidis JPA, Hemkens LG. Association of Convalescent Plasma Treatment With Clinical Outcomes in Patients With COVID-19: A Systematic Review and Meta-analysis. JAMA. 2021 Mar 23;325(12):1185-1195. doi: 10.1001/jama.2021.2747. PMID 33635310
- [Derived] Lovre D, Qadir MMF, Bateman K, Saltzman LY, Sherman M, Mauvais-Jarvis F. Acute estradiol and progesterone therapy in hospitalized adults to reduce COVID-19 severity: a randomized control trial. Sci Rep. 2024 Sep 30;14(1):22732. doi: 10.1038/s41598-024-73263-5. PMID 39349554
- [Derived] Ramanadhan S, Hansen K, Henderson JT, Cohen MA, Paynter R, Edelman A. Risk of thromboembolism in patients with COVID-19 who are using hormonal contraception. Cochrane Database Syst Rev. 2023 May 15;5(5):CD014908. doi: 10.1002/14651858.CD014908.pub3. PMID 37184292
- [Derived] Cohen MA, Edelman A, Paynter R, Henderson JT. Risk of thromboembolism in patients with COVID-19 who are using hormonal contraception. Cochrane Database Syst Rev. 2023 Jan 9;1(1):CD014908. doi: 10.1002/14651858.CD014908.pub2. PMID 36622724
- [Derived] Lovre D, Bateman K, Sherman M, Fonseca VA, Lefante J, Mauvais-Jarvis F. Acute estradiol and progesterone therapy in hospitalised adults to reduce COVID-19 severity: a randomised control trial. BMJ Open. 2021 Nov 30;11(11):e053684. doi: 10.1136/bmjopen-2021-053684. PMID 34848523

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol and Progesterone Arm: Standard of Care along with Estradiol Cypionate 5mg intramuscular injection at admission and Progesterone 200mg by mouth daily for 5 days starting at admission.
  Estradiol Cypionate 5 mg/ml: Standard of Care along with Estradiol Cypionate 5mg intramuscular injection at admission.
  Progesterone 200 mg Oral Capsule: Standard of Care along with Progesterone 200mg by mouth daily for 5 days starting at admission.
- Normal Saline and Folic Acid Arm: Standard of Care along with placebo-equivalent injection (1mL Normal Saline intramuscular injection) at admission and placebo-equivalent pill (folic acid 400 mg pill) daily for 5 days starting at admission.
  Standard of Care consistent with the National Institutes of Health (NIH) COVID-19 Treatment Guidelines.
  Placebo injection and placebo pill: Standard of Care consistent with the National Institutes of Health (NIH) Corona Virus Disease (COVID-19) Treatment Guidelines
Period: Overall Study
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Saline and Folic Acid Arm: Standard of Care along with placebo-equivalent injection (1mL Normal Saline intramuscular injection) at admission and placebo-equivalent pill (folic acid 400 mg pill) daily for 5 days starting at admission.
  Standard of Care consistent with the National Institutes of Health (NIH) COVID-19 Treatment Guidelines.
  Placebo injection and placebo pill: Standard of Care consistent with the National Institutes of Health (NIH) COVID-19 Treatment Guidelines
- Total: Total of all reporting groups
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (12.92) | 45.6 (13.41) | 48.5 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 24.5 (5.47) | 38.76 (6.87) | 31.63 (9.52)
Smoking status [Number; unit: partipants]
  Smokers | 4 | 2 | 6
  Non smokers | 1 | 3 | 4
Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] | 140.8 (18.21) | 139.4 (18.97) | 140.1 (17.54)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 91 (18) | 75.6 (14.76) | 83.3 (17.5)
Heart rate [Mean (Standard Deviation); unit: Beats per minute (Bpm)] | 94.2 (14.67) | 97.6 (10.19) | 95.9 (12.04)
O2 saturation [Mean (Standard Deviation); unit: Percentage of O2 saturation] | 93 (4.8) | 88.4 (5.18) | 90.7 (5.29)
Temperature [Mean (Standard Deviation); unit: Fahrenheit] | 98.38 (1.33) | 100.26 (1.07) | 99.32 (1.5)
World Health Organization (WHO) Score of 3 to 5 at randomization [Count of Participants; unit: Participants] — World Health Organization 9 point Ordinal Scale for Clinical Improvement in which lower score mean healthier participant. the score ranges from 0 to 8, 0 is uninfected, no clinical or virological evidence of infection, and 8 is dead, death. Study inclusion criteria was WHO score 3 to 5. Score 3 is participant hospitalized with mild disease and not on oxygen therapy. Score 4 is hospitalized with mild disease and is using oxygen by mask or nasal prongs. Score 5 is hospitalized with severe disease and on non-invasive ventilation or high-flow oxygen.
  Participants | 5 | 5 | 10
Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: Units/L] | 78.8 (74.97) | 78.2 (61.22) | 78.5 (64.53)
Alanine transaminase (ALT) [Mean (Standard Deviation); unit: Units/L] | 62.6 (60.01) | 70.2 (47.52) | 66.4 (51.19)
Neutrophil lymphocyte ratio (NLR) [Mean (Standard Deviation); unit: Ratio] | 3.96 (0.86) | 3.85 (2.61) | 3.90 (1.84)
White blood Cells (WBC) [Mean (Standard Deviation); unit: 10^9 cells per liter.] | 6.62 (0.72) | 6.38 (1.91) | 6.5 (1.37)
Platelet count [Mean (Standard Deviation); unit: 10^9 cells per liter] | 260 (66.49) | 157.8 (39.88) | 208.9 (74.65)
Charlson Comorbidity Index (CCI) [Mean (Standard Deviation); unit: units on a scale] — CCI is a chart review tool that quantifies an individual's burden of disease. The score is determined based on subject's age and medical conditions including Myocardial Infection, congestive heart failure, peripheral vascular disease, cerebrovascular accident or transient ischemic attack, etc. The lower the CCI score the less sick individual is and higher the score the more sick the individual. The minimum score is 0 if person is healthy and under 50 years of age and maximum score is 24 when an individual has all co-morbid conditions on the score list.
  units on a scale | 2.4 (1.82) | 1.4 (1.34) | 1.9 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Scores 1 or 2 on the 9-point World Health Organization (WHO) Ordinal Scale at Discharge, Measured up to Day 21
Description: The proportion will be calculated based on WHO ordinal scale for clinical improvement. The scale is from 0 to 8, with a higher score indicating worse clinical status.
  * Uninfected: No clinical or virological evidence of infection 0
  * Ambulatory: No limitation of activities 1 Limitation of activities 2
  * Hospitalized Mild Disease Hospitalized, no oxygen therapy 3 Oxygen by mask or nasal prongs 4
  * Hospitalized Severe Disease Non-invasive ventilation or high flow oxygen 5 Intubation and mechanical ventilation 6 Ventilation + additional organ support - 7 pressors, Renal Replacement Therapy (RRT), Extracorporeal Membrane Oxygenation (ECMO)
  * Dead Death 8
Time Frame: At discharge, measured up to Day 21
Population: Number of participants who achieved WHO score of 1 to 2 at discharge, measured up to Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
Participants | 5 | 4

2. Secondary Outcome: Length of Hospital Stay
Description: The investigators will review patients' medical records on day 14 and day 28. Then, the investigators will call patients on day 60. This will be done to determine the efficiency of treatment on length of hospital stay.
Time Frame: Baseline to day 60
Population: Medical records were reviewed at admission to day 60 to determine length of stay.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
Days | 7.2 (5.18) | 10.2 (7.53)

3. Secondary Outcome: Readmission
Description: The investigators will review patients' medical records on day 14 and day 28. Then, the investigators will call patients on day 60. This will be done to determine the readmission rates.
Time Frame: Baseline to day 60
Population: Medical records were reviewed from baseline to day 60 to determine readmission status
Measure: Number; unit: participants
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
participants
  COVID related readmission number | 0 | 0
  Non-COVID related readmission number | 0 | 1

4. Secondary Outcome: Number of Patients Requiring Invasive Mechanical Ventilation
Description: The investigators will review patients' medical records on day 14 and day 28. Then, the investigators will call patients on day 60. This will be done to determine the number of patients requiring invasive mechanical ventilation
Time Frame: Baseline to day 60
Population: Medical records were reviewed baseline to day 60 to determine number of patients requiring invasive mechanical ventilation
Measure: Number; unit: Participants
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
Participants | 0 | 1

5. Secondary Outcome: Number of Days Death Occurred After Admission
Description: The investigators will review patients' medical records on day 14 and day 28 and calculate number of deaths that occurred after admission. Then, the investigators will call patients on day 60. This will be done to determine the number of days death occurred after admission.
Time Frame: Baseline to day 60
Population: Medical records were reviewed from baseline to day 60 to determine the number of days death occurred after admission. One person died on day 19 after admission in the control arm.
Measure: Number; unit: Days
Arm/Group | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 1
Days | 19

6. Secondary Outcome: Number of Participants With Each Cause of Death
Description: The investigators will review patients' medical records on day 14 and day 28 and determine the cause of death. Then, the investigators will call patients on day 60. This will be done to determine the cause of death.
Time Frame: Baseline to day 60
Population: Medical records were reviewed from baseline to day 60 to determine the cause of death that occurred after admission for all 10 participants.
Measure: Number; unit: participants
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
participants
  Death from COVID-19 | 0 | 0
  Death from bacteremia | 0 | 1

7. Secondary Outcome: Grade 3 Adverse Events Occurrence
Description: Subjects will be followed daily for 7 days after initiation of treatment for adverse events. The investigators will review patients' medical records on day 14 and day 28. Then, the investigators will call patients on day 60. This will be done to determine the frequency and severity of adverse events in treatment arm vs. control arm.
Time Frame: Baseline to day 60
Population: Subjects were followed daily for 7 days after initiation of treatment for adverse events. Medical records were reviewed from baseline to day 60 to determine frequency and severity of adverse events in treatment arm vs. control arm.
Measure: Number; unit: Participants
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

8. Secondary Outcome: Serious Adverse Events Occurrence
Description: Subjects will be followed daily for 7 days after initiation of treatment for serious adverse events. The investigators will review patients' medical records on day 14 and day 28. Then, the investigators will call patients on day 60. This will be done to determine the frequency of serious adverse events in treatment arm vs. control arm.
Time Frame: Baseline to day 60
Population: Subjects were followed daily for 7 days after initiation of treatment for serious adverse events. Medical records were reviewed from baseline to day 60 to determine frequency of serious adverse events in treatment arm vs. control arm.
Measure: Number; unit: Participants
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
Number analyzed (Participants) | 5 | 5
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline to 60 days.
Arm/Group | Estradiol and Progesterone Arm | Normal Saline and Folic Acid Arm
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol and Progesterone Arm (N=5) | Normal Saline and Folic Acid Arm (N=5)
Death (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Bacteremia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol and Progesterone Arm (N=5) | Normal Saline and Folic Acid Arm (N=5)
Thrombophlebitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Bilateral upper cephalic basilic thrombophlebitis

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT04865029/Prot_SAP_000.pdf